CLINICAL TRIAL: NCT06855459
Title: A Randomized Double Blinded and Placebo-Controlled Trial to Assess the Impact of Biophoton Therapy on Self-Grown Stem Cells
Brief Title: The Impact of Biophoton Therapy on Self-Grown Stem Cells
Acronym: Stem Cells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Institute of All Medicines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FIAM-SC255
Record Dates: First submitted 2025-02-26; First posted 2025-03-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Increase the Total Number of Stem Cells; Inflammation
Keywords: Biophoton Therapy, Tesla BioHealing, Stem Cells; Increase Stem Cells
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, placebo-controlled intervention clinical study to assess the effectiveness of biophoton therapy in impacting stem cells. Approximately 46 volunteers who want to increase self-grown stem cells will participate in the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each set of the study device is labelled with a unique code for use by only one participant. Participant, investigator data analyzer are all blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): This arm is to verify if biophoton generators can increase self-grown stem cells as previously observed that using Tesla BioHealers for 2 weeks the self-grown stem cells increased by 346%. BioHealing Biophotonizer-A had been used to increase is an over-the-counter (OTC) medical device and it can be used by anyone who wants to increase blood circulation and reduce bodily pains. For this study, the active Biophotonizer-A will be labeled with a code. The participant cannot know if the devices are active or inactive. When the participant places the devices close to the body, she/he may or may not receive life force energy. The participant will record changes in pain, quality of life at baseline and at the end of each week. A total of 23 participants will be enrolled in this group.
  Interventions: Device: Biophoton Generators
- Placebo Control (Placebo Comparator): Each participant assigned to the Control Group will be treated with the 4 placebo devices
  Interventions: Device: Biophoton Generators

INTERVENTIONS:
Device: Biophoton Generators — Users will be receiving biophotons emitted from the 4 devices during sleep and other time.

SUMMARY:
Study Objective The purpose of this clinical study is to evaluate if biophoton therapy, delivered by Tesla BioHealing® Biophoton Generators (Biophotonizer), can increase self-grown stem cells naturally.

Study Design This is a randomized, double-blinded, placebo-controlled intervention clinical study to assess the effectiveness of biophoton therapy in impacting stem cells. Approximately 46 volunteers who want to increase self-grown stem cells will participate in the study.

Study Randomization The biostatistician will prepare a randomization schedule including a serial of subject numbers. A subject number will be randomly assigned to each study participant, which will assign them to either the control group or the treatment group.

Other than the Informed Consent Form (ICF), all study information will be recorded by using the subject number. The Principal Investigator, study physicians, study nurse, data-entry specialists, and biostatisticians, as well as the participants, will be blinded about who received which product during the first two weeks of study participation.

DETAILED DESCRIPTION:
Study Enrollment Each potentially qualified volunteer will review the Informed Consent Form online (e-ICF) and Enrollment Criteria online (e-Criteria) first, then discuss the e-ICF and e-Criteria with the study team medical professional via telephone during the scheduled time. Each qualified volunteer will sign the e-ICF and send it to the Medical Office Coordinator. The Coordinator will assign the qualified volunteer a randomized subject number, then the volunteer will become a study participant.

Study Procedure We expect that the participant will stay in this clinical treatment for 2 weeks, or 4 weeks if the participants are randomly placed in a placebo group. The first 2 weeks of participation are double blinded to record the placebo effects, as each set of the study device is labelled with a unique code for use by only one participant. The change of the placebo device to the treatment device will be performed by the study device management team staff who will not inform the study participant nor study research staff who involve study data collection. Each participant assigned to the Control Group will be treated with the 4 placebo devices and placed on the 4 corners of the bed. Each participant assigned to the Treatment Group will receive 4 Biophoton generator devices and placed on the 4 corners of the bed. Each participant will use the Treatment or Control device for at least 8 hours every night for the 2 weeks during sleep. During the day, participants are welcome to bring the study devices and place them near the body during the daytime. At the end of the initial 2 weeks, study participants randomized to the Placebo group will be advised whether they will use the Open-Labeled product to treat them for 2 weeks. Each participant will be guided by study team staff to perform the following tests on their assigned testing days: a visual analog scale of pain, the standard SF-36 questionnaires (SF-36) for measuring life quality, and stem cell examination respectively at the Baseline, one and two weeks after using the study devices.

Study Supply All study devices (Placebo or Treatment) will be packed for easy use. Each participant will use the assigned devices during the 2-week study period (Treatment Group), or for 2+2 weeks (Placebo Group) after being switched to the Treatment group after the first two weeks of the placebo period.

Study Patient Population The adult who wants to increase stem cells without major health issues.

Investigational Product and Mode of Administration Tesla BioHealing Biophotonizer-A is an over-the-counter (OTC) medical device and it can be used by anyone who wants to increase blood circulation and reduce bodily pains. For this study, the active or inactive Biophotonizer-A will be labeled with a code. The participant and/or caregiver cannot know if the devices are active or inactive. When the participant places the devices close to the body, she/he may or may not receive life force energy. The participant will record changes in pain, quality of life at baseline and at the end of each week.

Comparator and Mode of Administration Clinical measurements will be conducted by medical professionals. The same shape, size, and weight of the device without generating biophoton is to be labeled with a random code and used as a comparator. The comparator device will be placed at the 4 corners of the bed during nightly sleep during the entire study period. The participant will record the life quality changes and answer the 10-point pain scale questionnaires. Clinical measurements will be conducted by medical professionals.

Study Duration Estimated date of the first patient enrolled: January 14, 2025. The estimated date of the last participant completed: December 15, 2025.

Duration of Treatment Participants in the Treatment Group and Control Group will actively participate in the study for 2 or 4 weeks. Each Participant will answer the standard study questionnaires respectively at the baseline, at the end of each week.

If the participant wants to continually improve her/his stem cell counts after completing the study, the active device can be continually used for four more weeks with a small rental fee. Then, all study devices will be shipped back to the study center.

Outcome Variables

Primary Outcome Measure:

Stem cell counts. [Time Frame: baseline, 0-2, 0-4 weeks].

Secondary Outcome Measure:

1. Life Quality. Short Form Health Survey (SF-36) [Time Frame: baseline, 0-1, 0-2, 0-3, 0-4, is to measure the quality of life as influenced by the investigational medical device. SF-36 has been used worldwide as a standard clinical research tool.
2. Pain Disability Index (PDI) [Time Frame: baseline, 0-1, 0-2, 0-3, 0-4]. The PDI measures the degree to which pain impacts 7 different categories of daily activities.
3. Pain medicine use. The reported pain medicine use will be tabulated and analyzed. [Time Frame: baseline, 0-1, 0-2, 0-3, 0-4].

Safety Outcome: Occurrence of adverse events. Any adverse events were reported by participants. [Time Frame: Any Adverse Events occurred at the baseline, and up to 4 weeks.] Any adverse events reported by participants will be tabulated and compared between the two groups.

Eligibility Criteria

Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial.
* Is able and willing to comply with all trial requirements.
* Male or female ages 18-70 years old without major diseases.
* Participants must not be heavy users of Tesla BioHealing devices; enrollment will be determined by the clinical team based on an evaluation of the participant's prior device usage.
* Must be fluent in English.

Exclusion Criteria:

* Untreated psychiatric disturbances that would affect trial participation as judged by the research medical professional.
* Is participating in another investigational drug or device trial
* Had been treated with Stem Cell therapy within a 6-month period.

Statistical Methods The sample size is calculated based on the primary efficacy variable and the data from the pilot study in self-grown stem cells (more than 70% success, for the treatment, and less than 10% success for the not treated) to compare the treatment with Biophoton Generator, which was at least 70% successful and to compare with placebo.

We plan to enroll 23 Participants in each group to have 19 completers by adding 4 (20%) more participants. Therefore, a total of 46 participants will be enrolled. If the Principal Investigator decides to increase the enrolment to enable statistical difference between the two groups, the enrollment can be continual. Primary and secondary outcome variables will be statistically analyzed by using Chi-square analysis or paired T-Test.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial.
* Is able and willing to comply with all trial requirements.
* Male or female ages 18-70 years old without major diseases.
* Participants must not be heavy users of Tesla BioHealing devices; enrollment will be determined by the clinical team based on an evaluation of the participant's prior device usage.
* Must be fluent in English.

Exclusion Criteria:

* Untreated psychiatric disturbances that would affect trial participation as judged by the research medical professional.
* Is participating in another investigational drug or device trial
* Had been treated with Stem Cell therapy within a 6-month period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Self-Grown Stem Cells Count | [Time Frame: baseline, 0-2, 0-4 weeks].
  To determine if treatment with Biophoton Generator can impact self-grown steam cells naturally

SECONDARY OUTCOMES:
Quality of Life Short Form -36 (SF-36) -the function and well-being of a person | [Time Frame: baseline, 0-2, 0-4 weeks].
  To determine if treatment with Biophoton Generator can significantly improve life quality. The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status.
Impact of Biophoton Treatment on Pain Disability Index | [Time Frame: baseline, 0-2, 0-4 weeks].
  To determine if treatment with a Biophoton Generator can improve the ability to complete daily life activities. The rating scales are designed to measure the degree to which aspects of your life are disrupted by chronic pain. For each of the 7 categories of life activity listed, please circle the number on the scale that describes the level of disability you typically experience. A score of 0 means no disability at all, and a score of 10 signifies that all of the activities in which you would normally be involved have been disrupted or prevented by the pain.

CONTACTS AND LOCATIONS:
Overall Officials: James Z Liu, MD, PhD, Study Chair — First Institute of All Medicines
Locations (2):
- United States (2):
  - Tesla MedBed at Tampa-FL, Tampa, Florida
  - Tesla BioHealing Wellness Hotel - Butler-PA, Butler, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Plan for Sharing Individual Participant Data (IPD)
  * Data Sharing Statement: IPD will be shared as de-identified data, including study protocol, statistical analysis plan, informed consent form, and clinical study report.
  * Timeframe: Data will be available within 6-12 months after publication and accessible for at least 5 years.
  * Data Access: Stored in ClinicalTrials.gov, Vivli, or Dryad, data will be shared upon formal request with a research proposal. Requests will be reviewed by a Data Access Committee (DAC) based on scientific validity and ethical compliance.
  * Privacy Protection: Data will be anonymized per HIPAA/GDPR standards, ensuring participant confidentiality.
  * Usage: Available for meta-analyses and secondary research, with proper citation required. Commercial use is prohibited.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The anticipated availability period will be within 6 to 12 months after publication.
Access Criteria: Data will be stored in a secure, recognized repository such as ClinicalTrials.gov
URL: http://www/firstallmed.org